CLINICAL TRIAL: NCT00856661
Title: A Randomised, Double-Blind, Parallel-Group Placebo-Controlled Phase III Study to Evaluate the Efficacy and Safety of Desmoteplase in Subjects With Acute Ischemic Stroke
Brief Title: Efficacy and Safety Study of Desmoteplase to Treat Acute Ischemic Stroke (DIAS-4)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The recruitment into DIAS4 has been stopped as the result of DIAS 3 indicates that the study is unlikely to reach its primary endpoint with the current protocol
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12649A; 2008-005539-14 (EudraCT Number)
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Stroke
Keywords: Acute ischemic stroke; Angiography; Desmoteplase; Thrombolytic
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — salivary plasminogen activator alpha 1, Desmodus rotundus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desmoteplase (Experimental)
  Interventions: Drug: Desmoteplase
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmoteplase — 90 μg/kg bodyweight, IV, single bolus over 1 to 2 minutes on 1st day
  Arms: Desmoteplase
Drug: Placebo — IV, single bolus over 1 to 2 minutes on 1st day
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether desmoteplase is effective and safe in the treatment of patients with acute ischaemic stroke when given within 3 to 9 hours from onset of stroke symptoms.

DETAILED DESCRIPTION:
Acute stroke is a major cause of mortality and long-term disability in the developed world. The only currently approved thrombolytic intervention for acute ischemic stroke, which constitutes the majority of strokes, is alteplase (recombinant tissue plasminogen activator; rtPA). The use of alteplase is limited as it is approved for use within 3 hours after symptom onset and by the risk of inducing intracerebral haemorrhage; consequently fewer than 3% of acute stroke subjects are treated. The thrombolytic agent desmoteplase (recombinant Desmodus Salivary Plasminogen Activator alpha-1; rDSPAalpha-1) produced by recombinant biotechnology has its naturally occurring counterpart in the saliva of the vampire bat Desmodus rotundus. Compared to alteplase, desmoteplase has a more favourable profile in terms of high fibrin specificity and non neurotoxicity.

The study aims to confirm efficacy and safety of desmoteplase for thrombolytic therapy of patients with acute ischaemic stroke in the extended time window of 3 to 9 hours after onset of stroke symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute ischemic stroke
* Informed consent
* Age between 18 and 85 years
* Treatment can be initiated within 3 to 9 hours after the onset of stroke symptoms
* NIHSS Score of 4 to 24
* Vessel occlusion or high-grade stenosis on MRI or CTA in proximal cerebral arteries

Exclusion Criteria:

* Pre-stroke mRS >1
* Previous exposure to desmoteplase
* Extensive early infarction on MRI or CT in any affected area
* Imaging evidence of ICH or SAH; AV malformation; cerebral aneurysm; or cerebral neoplasm
* Internal carotid artery occlusion on the side of the stroke lesion
* Treatment with heparin in the past 48 hours and a prolonged partial thromboplastin time
* Treatment with oral anticoagulants and a prolonged prothrombin time
* Treatment with glycoprotein IIb - IIIa inhibitors within the past 72 hours. Use of single agent oral platelet inhibitors is permitted
* Treatment with a thrombolytic agent within the past 72 hours

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2009-04; Primary Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (152):
- United States (81):
  - US053, Phoenix, Arizona
  - US081, Castro Valley, California
  - US089, La Jolla, California
  - US043, Loma Linda, California
  - US008, Los Angeles, California
  - US020, Palo Alto, California
  - US050, Pasadena, California
  - US098, Santa Barbara, California
  - US051, Thousand Oaks, California
  - US068, Englewood, Colorado
  - US063, Fairfield, Connecticut
  - US104, New Haven, Connecticut
  - US049, Pensacola, Florida
  - US109, Atlanta, Georgia
  - US042, Augusta, Georgia
  - US052, Columbus, Georgia
  - US080, Decatur, Georgia
  - US040, Lawrenceville, Georgia
  - US067, Macon, Georgia
  - US085, Savannah, Georgia
  - US086, Savannah, Georgia
  - US093, Chicago, Illinois
  - US101, Chicago, Illinois
  - US044, Chicago, Illinois
  - US074, Evanston, Illinois
  - US073, Glenview, Illinois
  - US091, Maywood, Illinois
  - US088, Oak Lawn, Illinois
  - US016, Indianapolis, Indiana
  - US072, Des Moines, Iowa
  - US061, New Orleans, Louisiana
  - US108, New Orleans, Louisiana
  - US064, Shreveport, Louisiana
  - US014, Baltimore, Maryland
  - US039, Boston, Massachusetts
  - US003, Boston, Massachusetts
  - US017, Worcester, Massachusetts
  - US066, Detroit, Michigan
  - US096, Detroit, Michigan
  - US083, Detroit, Michigan
  - US060, Grand Blanc, Michigan
  - US078, Grand Rapids, Michigan
  - US103, Kalamazoo, Michigan
  - US056, Petoskey, Michigan
  - US113, Royal Oak, Michigan
  - US076, Southfield, Michigan
  - US082, Southfield, Michigan
  - US079, Troy, Michigan
  - US059, Gulfport, Mississippi
  - US048, Springfield, Missouri
  - US077, Lebanon, New Hampshire
  - US055, Edison, New Jersey
  - US115, Neptune City, New Jersey
  - US100, Ridgewood, New Jersey
  - US075, Albany, New York
  - US102, Brooklyn, New York
  - US012, Buffalo, New York
  - US026, Stony Brook, New York
  - US037, Greensboro, North Carolina
  - US069, Winston-Salem, North Carolina
  - US038, Cleveland, Ohio
  - US001, Columbus, Ohio
  - US062, Columbus, Ohio
  - US046, Toledo, Ohio
  - US095, Springfield, Oregon
  - US070, Allentown, Pennsylvania
  - US023, Philadelphia, Pennsylvania
  - US099, Pittsburgh, Pennsylvania
  - US084, Pittsburgh, Pennsylvania
  - US092, Providence, Rhode Island
  - US087, Warwick, Rhode Island
  - US057, Columbia, South Carolina
  - US019, Chattanooga, Tennessee
  - US058, Nashville, Tennessee
  - US021, Houston, Texas
  - US031, Houston, Texas
  - US112, Houston, Texas
  - US047, Richmond, Virginia
  - US006, Winchester, Virginia
  - US011, Madison, Wisconsin
  - US097, Milwaukee, Wisconsin
- Belgium (4):
  - BE008, Bruges
  - BE004, Hasselt
  - BE005, Roeselare
  - BE006, Wilrijk
- Brazil (7):
  - BR012, Campinas
  - BR004, Porto Alegre
  - BR008, Porto Alegre
  - BR007, Porto Alegre
  - BR009, Rio de Janeiro
  - BR011, Rio de Janeiro
  - BR006, Salvador
- Canada (8):
  - CA001, Calgary, Alberta
  - CA004, Edmonton
  - CA006, Halifax
  - CA008, Mississauga
  - CA007, Ottawa
  - CA012, Toronto
  - CA002, Toronto
  - CA005, Victoria
- Chile (5):
  - CL002, Santiago
  - CL003, Santiago
  - CL004, Santiago
  - CL006, Santiago
  - CL005, Valparaíso
- Denmark (4):
  - DK002, Aalborg
  - DK001, Aarhus
  - DK004, Copenhagen NV
  - DK003, Glostrup Municipality
- Finland (3):
  - FI001, Helsinki
  - FI002, Tampere
  - FI003, Turku
- IE001, Dublin, Ireland
- Italy (12):
  - IT010, Ancona
  - IT008, Brescia
  - IT003, Florence
  - IT004, Imperia
  - IT002, Milan
  - IT006, Milan
  - IT009, Milan
  - IT012, Modena
  - IT001, Rome
  - IT005, Rome
  - IT007, Rozzano
  - IT011, Verona
- Mexico (4):
  - MX002, D.f.
  - MX003, Mexico City
  - MX004, Mexico City
  - MX005, Monterrey Nuevo Leon
- Norway (3):
  - NO003, Bergen
  - NO001, Oslo
  - NO002, Trondheim
- South Africa (3):
  - ZA003, Cape Town
  - ZA002, Cape Town
  - ZA001, Cape Town
- Sweden (2):
  - SE002, Lund
  - SE001, Malmo
- United Kingdom (15):
  - GB012, Belfast
  - GB004, Christchurch
  - GB010, Dundee
  - GB002, Exeter
  - GB009, Glasgow
  - GB007, Glasgow
  - GB011, Liverpool
  - GB006, London
  - GB003, London
  - GB001, Newcastle upon Tyne
  - GB016, Nottingham
  - GB014, Sheffield
  - GB005, Stoke-on-Trent
  - GB015, Westcliff-on-Sea
  - GB013, Wolverhampton

REFERENCES:
- [Derived] von Kummer R, Mori E, Truelsen T, Jensen JS, Gronning BA, Fiebach JB, Lovblad KO, Pedraza S, Romero JM, Chabriat H, Chang KC, Davalos A, Ford GA, Grotta J, Kaste M, Schwamm LH, Shuaib A, Albers GW; DIAS-4 Investigators. Desmoteplase 3 to 9 Hours After Major Artery Occlusion Stroke: The DIAS-4 Trial (Efficacy and Safety Study of Desmoteplase to Treat Acute Ischemic Stroke). Stroke. 2016 Dec;47(12):2880-2887. doi: 10.1161/STROKEAHA.116.013715. Epub 2016 Nov 1. PMID 27803391
- See also: EMA EudraCT Results: 2008-005539-14 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2008-005539-14/results

RESULTS

PARTICIPANT FLOW:
Groups:
- Desmoteplase: 90 μg/kg bodyweight, IV, single bolus over 1 to 2 minutes 3-9 hours after symptoms onset
- Placebo: Placebo: IV, single bolus over 1 to 2 minutes 3-9 hours after symptoms onset
Period: Overall Study
Arm/Group | Desmoteplase | Placebo
Started | 135 (Randomised) | 135 (Randomised)
Treated | 126 | 131
Randomized Not Treated | 9 | 4
Completed | 108 | 106
Not Completed | 27 | 29
Not completed — Death | 15 | 18
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Judgement | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Desmoteplase: Desmoteplase: 90 μg/kg bodyweight, IV, single bolus over 1 to 2 minutes 3-9 hours after symptoms onset
- Total: Total of all reporting groups
Arm/Group | Desmoteplase | Placebo | Total
Number analyzed (Participants) | 135 | 135 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (11.1) | 68.2 (12.5) | 68.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 69 | 141
  Male | 63 | 66 | 129
Race/Ethnicity, Customized [Number; unit: participants]
  White | 111 | 115 | 226
  Black or african americal | 11 | 9 | 20
  Asian | 7 | 6 | 13
  Other | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Modified Rankin Scale Score (mRS) (Percentage of Participants With mRS Scores 0-2)
Description: The mRS is a clinician-rated scale designed to provide a global assessment of the patients dependency after stroke. The scale consists of a single item measuring the patient's function based on the ability to perform daily activities. The patient is rated on a 7-point scale from 0 to 6, where a score of 5 corresponds to severe disability, and 6 to death. Assessment of a pre-stroke mRS score is based on an interview addressing the status of the patient prior to the stroke
Time Frame: Day 90
Population: Two and three patients from the desmoteplase and placebo group, respectively, had no valid functional assessment done. Hence, the full analysis set consisted of 124 and 128 patients, respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | Desmoteplase | Placebo
Number analyzed (Participants) | 124 | 128
Percentage of participants | 41.9 | 35.9
Statistical Analysis 1: Comparison: Desmoteplase vs Placebo; All patients who were treated and had at least one valid post-baseline assessment of the mRS. As death is a valid outcome on the mRS, patients who died within 90 days after IMP administration were included; Test type: Superiority or Other; p = 0.2290, Regression, Logistic; If no assessment was available for last observation carried forward after baseline, the mRS score was set to 5 if alive, or 6, if otherwise = death; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.79 to 2.64]

2. Secondary Outcome: National Institutes of Health Stroke Scale (NIHSS) Score. (Percentage of Participants With NIHSS Scores <=1 or NIHSS Decrease >=8)
Description: The NIHSS is a clinician-rated, 15-item scale designed to assess the severity of stroke-related neurological deficits: level of consciousness, eye movements, visual fields, facial symmetry, motor strength (arm and leg), coordination, sensation, language (aphasia and dysarthria), and neglect. Each item is rated on a 3-, 4-, or 5-point scale ranging from 0 (normal) to the maximum score (extremely severe symptoms). The total score of the 15 items ranges from 0 to 42, where lower scores indicate less impairment.
Time Frame: 90 days
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Desmoteplase | Placebo
Number analyzed (Participants) | 124 | 128
Percentage of participants | 49.2 | 50.8
Statistical Analysis 1: Comparison: Desmoteplase vs Placebo; Test type: Superiority or Other; p = 0.9401, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.59 to 1.62]

3. Secondary Outcome: Composite of mRS & NIHSS Response (Percentage of Participants With mRS Scores 0-2 and (NIHSS <= 1 or NIHSS Decrease >= 8)
Description: Please see outcomes measure one and two for detailed description of the scales
Time Frame: Day 90
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Desmoteplase | Placebo
Number analyzed (Participants) | 124 | 128
Percentage of participants | 32.3 | 28.9
Statistical Analysis 1: Comparison: Desmoteplase vs Placebo; All patients treated, who had at least one valid post-baseline assessment of the mRS and with a baseline NIHSS score of 8 to 24. If no assessment was available for last observation carried forward after baseline, the mRS score was set to 5 if the patient was known to be alive, or 6, if otherwise = dead; Test type: Superiority or Other; p = 0.5076, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.68 to 2.18]

4. Secondary Outcome: Modified Ranking Scale Score (Using the Ordinal Scale)
Description: Please see outcomes measure one for detailed description of the mRS scale
Time Frame: Day 90
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Desmoteplase | Placebo
Number analyzed (Participants) | 124 | 128
Scores on a scale | 3.02 (0.14) | 3.12 (0.15)
Statistical Analysis 1: Comparison: Desmoteplase vs Placebo; all patients treated, who had at least one valid post-baseline assessment of the mRS. As death is a valid outcome on the mRS, patients who died within 90 days after IMP administration were included; Test type: Superiority or Other; p = 0.6146, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.72 to 1.75]

ADVERSE EVENTS:
Time Frame: baseline to end of study
Groups:
- Desmoteplase: Desmoteplase: 90 ug/kg, IV, single bolus over 1 to 2 minutes 3-9 hours after symptoms onset
Arm/Group | Placebo | Desmoteplase
Serious Adverse Events (participants affected / at risk) | 56/131 | 61/126
Other Adverse Events (participants affected / at risk) | 107/131 | 98/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=131) | Desmoteplase (N=126)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 4 | 4
Bradycardia (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Pupils unequal (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Catheter site phlebitis (General disorders) | 0 | 1
Death (General disorders) | 0 | 1 — Deaths after end of study (day 167). Only deaths occuring within 90 days of IMP are reported in main study
Multi-organ failure (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 3
Pneumonia bacterial (Infections and infestations) | 4 | 5
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood culture positive (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 4 | 2
Nih stroke scale score increased (Investigations) | 4 | 0
Oxygen saturation decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Respiratory rate increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 6 | 3
Brain stem stroke (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 2
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 4
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 5 | 3
Loss of consciousness (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 2 | 0
Stroke in evolution (Nervous system disorders) | 6 | 10
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 3
Agitation (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=131) | Desmoteplase (N=126)
Atrial fibrillation (Cardiac disorders) | 13 | 11
Constipation (Gastrointestinal disorders) | 32 | 30
Diarrhoea (Gastrointestinal disorders) | 8 | 6
Nausea (Gastrointestinal disorders) | 14 | 12
Vomiting (Gastrointestinal disorders) | 13 | 7
Oedema peripheral (General disorders) | 1 | 11
Pain (General disorders) | 7 | 7
Pyrexia (General disorders) | 11 | 8
Pneumonia bacterial (Infections and infestations) | 7 | 3
Urinary tract infection (Infections and infestations) | 4 | 8
Urinary tract infection bacterial (Infections and infestations) | 26 | 22
Fall (Injury, poisoning and procedural complications) | 9 | 3
Blood potassium decreased (Investigations) | 4 | 8
Nih stroke scale score increased (Investigations) | 10 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 12 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 9
Headache (Nervous system disorders) | 22 | 22
Stroke in evolution (Nervous system disorders) | 7 | 7
Anxiety (Psychiatric disorders) | 8 | 11
Depressive symptom (Psychiatric disorders) | 13 | 13
Insomnia (Psychiatric disorders) | 11 | 15
Haematuria (Renal and urinary disorders) | 7 | 6
Urinary retention (Renal and urinary disorders) | 8 | 3
Hypertension (Vascular disorders) | 14 | 16
Hypotension (Vascular disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No